CLINICAL TRIAL: NCT04072718
Title: A Phase II Study of Simultaneous Integrated Boost With Volumetric Arc Radiotherapy After Breast Conservative Surgery in Patients With Breast Cancer
Brief Title: Simultaneous Integrated Boost With Volumetric Arc Radiotherapy in Patients With Breast Cancer
Acronym: SIBART-BC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2017/127
Record Dates: First submitted 2017-10-30; First posted 2019-08-28 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: Hypofractioned radiotherapy; Simultaneous integrated boost
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: To be treated with hypofractionated radiotherapy of 34Gy in 10 fractions to whole breast and 40Gy in 10fractions to the tumor bed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 34 Gy/10#/2wk to the PTV and 40Gy/10#/2 Wk to the PTV SIB with IGRT using Rapid arc technique.

SUMMARY:
The study will include 27 patients to study the dosimetric data and acute toxicity. Patients will be treated by SIB intensity modulated radiotherapy (IMRT) boost to the cavity.The dose to be delivered will be a hypo fractionated regimen of 34Gy/10#/2weeks to the whole breast and 40Gy/10#/2weeks to the tumour bed. The dose to the target and to the OAR will be observed. The acute toxicity and cosmesis will be assessed.

DETAILED DESCRIPTION:
Aim To study the dose to the target and OARs with SIB-IMRT in patients with breast cancer.

Objectives: To study

1. Dose distribution, target coverage and dose homogeneity in the diseased breast.
2. Dose to the OARs.
3. Acute toxicities.
4. Cosmetic outcome. Materials and methods Patients: Total 27 patients post BCS will be included in the study. 4D computed tomography simulation and image acquisition: All the patients will undergo a standard free breathing with virtual CT breast simulationin supine position on a breast board or wing board with ipsilateral arm abducted above head. The other side arm will be kept on side. Three skin markings will be placed along with the fiducials below the breast folds for reproducibility and the localizationtion of tumor bed. The 4DCT images with recording the respiratory signals will be acquired with thickness of 3mm with a 16 slice Brilliance 85cms bore CT scanner (Philips medical system, Inc., Cleveland, OH, USA). The signals will be sent to the scanner to label a time tag on each CT image. 4D software (GE Healthcare, Waukesha, WT, USA) will sort the reconstructed 4DCT image into ten separate phases on basis of these tags, with 0% corresponding to end-inhalation (CT0) and 50% corresponding to end-exhalation CT50. The constructed 4DCT sets will be transferred to eclipse treatment planning system (TPS), (Eclipse 10, Varian medical system, Palo alto, CA, USA) for structure delineation. The 10 to 90% phase of 4DCT images will be registered on 50% phase images, which will serve as basic phase image. The delineation of the tumor cavity and contouring of the organs at risk will be done by using standard RTOG guidelines for contouring breast cancer cases on Maximum intensity phase (MIP) CT. The tumor cavity will be delineated with the help of surgical clips (if put by the surgeon during lumpectomy), mammography films and by the clinical examination done before surgery to assess the location of tumor in the affected breast. The scar will be adequately covered. The organs at risk contoured will be heart, bilateral lungs, contralateral breast, esophagus, spinal cord, bilateral humerus head, left anterior descending(LAD) artery and right coronary artery. The diseased breast contoured will be clinical target volume (CTV). A margin of 5mm will be added for setup error and motion for the planning treatment volume (PTV) breast. A Margin of 5mm will be added to cavity to form PTV SIB.

Target coverage and dose homogeneity: target implies to the tumor bed which has been delineated with the help of surgical clips, mammography and clinical examination and history. It has to be covered adequately and the dose has to be homogenized without the presence of any cold spot or hotspot. The criteria to ensure the dose distribution appropriately will beas: PTV: D98 > 95% and D2 < 107%; PTV SIB: D98 > 95% and D2 < 107%. Dose to the OARs: OARs will include: heart, ipsilateral lung, contralateral lung, opposite breast, oesophagus, spinal cord and LAD. The dose constraints will be different to the laterality of the disease since the location of organs differs.

Treatment:Patients will be treated with a dose of 34 Gy/10#/2wk to the PTV and 40Gy/10#/2 Wk to the PTV SIB with IGRT using Rapid arc technique. Acute toxicities will be assessed at the time of completion of treatment andat 1 month and 3 months after treatment. Cosmetic outcome will be assessed at 1, 3 and at 6 months of followup.

Assessment of toxicity will be done as per RTOG scores and LENT SOMA scale Toxicity Grade0 Grade1 Grade2 Grade3 Grade4 Skin No change over baseline Follicular, faint/ dull erythema/ epilation/dry desquamation/ decreased sweating Tender or bright erythema, patchy moist desquamation/ moderate edema Confluent, moist desquamation other than skin folds, pitting edema Ulceration, haemorrhage, necrosis Subcutaneous tissue None Slight induration (fibrosis) and loss of subcutaneous fat Moderate fibrosis but asymptomatic Slight field contracture <10% linear reduction Severe induration and loss of subcutaneous tissue Field contracture >10% linear measurement Necrosis

Pigmentary change :

0 = None

1 = Transitory , slight 2 = Permanent , marked

Breast edema :

0 = None 1 = Asymptomatic 2 = Symptomatic 3 = Secondary dysfunction Cosmetic assessment Sample size calculation

The purpose of the trial is to reject the experimental treatment from further study if it were insufficiently active, and to accept it for further study if it were active. The study is designed as a phase II trial with the following assumptions:

* the inactivity cut-off is chosen equal to 11%, the activity cut-off equal to 36%. Hence the hypotheses of interest are H0: r ≤ 11% against HA: r ≥ 36%, where r is the proportion of patients with grade 2 skin toxicity
* the type I error rate (alpha, probability of accepting an overly toxic treatment, a false positive outcome) is set to 5%
* the type II error rate (beta, probability of rejecting an acceptably toxic treatment, a false negative outcome) is set to 10% - i.e., the power is equal to 90% Under these assumptions, the design consists of treating 27 evaluable patients, and if at most 5 patients have grade 2 skin toxicity, the treatment is considered acceptable (5/27=19%)
* if at least 6 patients have grade 2 skin toxicity, the treatment is considered too toxic (6/27=22%)

Statistical analysis The principle end point of the study will be an analysis of dosimetric parameters and acute radiation toxicities. Secondary end point will be cosmetic score analysis and local control. Skin, subcutaneous toxicity and cosmetic assessment will be done before treatment and then in regular follow up of the study. Descriptive statistics including mean and standard deviation will be obtained for all variables. p values of <0.05 will be taken as significant. All tests would be performed using SPSS (Statistical Package for the Social Sciences) v.12.0.

ELIGIBILITY:
Inclusion Criteria:

* Primary cancer of breast of any histology,
* age 18-60 years,
* post BCS,
* KPS >70,
* no distant metastasis and patients who have or have not received chemotherapy

Exclusion Criteria:

* History of prior primary malignancy,
* prior irradiation to breast or chest,
* pregnant or lactating women, and
* collagen vascular disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 27 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Acute radiation toxicities | one month after completion of treatment
  Acute skin toxicities will be assessed using RTOG acute toxicity scoring scale after one month of completion of treatment.

SECONDARY OUTCOMES:
cosmetic score analysis | 6 months, 1 year and 3 years off follow up.
  NSABP/HARVARD/RTOG criteria
  Pigmentary change :
  0 = None
  1 = Transitory , slight 2 = Permanent , marked
  Breast edema :
  0 = None 1 = Asymptomatic 2 = Symptomatic 3 = Secondary dysfunction
local control | 3 years
  Any recurrence in the involved breast.
Late toxicity | 3 years
  Late toxicities will be recorded and after treatment according to RTOG radiation morbidity scoring criteria

CONTACTS AND LOCATIONS:
Overall Officials: Budhi S Yadav, MD, Principal Investigator — Postgraduate Institute of Medical Education & Research
Locations (1):
- Dr Budhi Singh Yadav, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Acute Toxicity, dosimetry
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At 2 years and will be available till 5 years
Access Criteria: online